CLINICAL TRIAL: NCT05199857
Title: WE BEAT - HEART Club Fontan Wellness Project: A Virtual Resilience Promotion and Frailty Prevention Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Reuben Phoenix Schostak Fontan Wellness Project Fund (Unknown)
Responsible Party: Principal Investigator, Jesse Hansen, Assistant Professor of Pediatrics, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00205931
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Fontan Physiology; Frailty; Single Ventricle Heart Disease
Keywords: Wellness education; Exercise program
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellness education and Home exercise programs (Experimental)
  Interventions: Behavioral: WE BEAT Group Wellness Education program - phase 1; Behavioral: HEART Club Home Exercise program - phase 2

INTERVENTIONS:
Behavioral: WE BEAT Group Wellness Education program - phase 1 — Participants will be assigned into a small group with 3-6 other participants and will participate in a weekly, 45-50 minute intervention session for 5 weeks, delivered by a licensed clinical psychologist or limited licensed clinical psychology fellow using University of Michigan (UM) Zoom. Each session will focus on a particular skill related to wellness and resiliency. There will also be a short battery of questionnaires to complete.
Behavioral: HEART Club Home Exercise program - phase 2 — This is an individualized home exercise program adapted from the exercise programs used in traditional, hospital-based cardiac rehabilitation. A complete cardiopulmonary exercise test (CPET) may be completed if needed for a baseline and one will be done at the last visit. The exercise physiology team will discuss participants exercise goals, interests, and available resources to help develop the exercise plan for the research study. Once the program is designed, participants will complete the exercise activities in the plan. Over time, participants will advance through various stages in the program and then will be gradually introduced to the principles of exercise rehabilitation and more intense physical exercise. Participants will be asked to wear a wearable activity tracker and have scheduled video check-ins with the exercise physiology team. Throughout the program participants will complete a short battery of surveys.

SUMMARY:
This trial is being conducted to evaluate the effect of a small-group wellness education program combined with a longitudinal, individualized prescription exercise program on the wellness, resiliency, and daily activity levels of pediatric patients with Fontan physiology.

There will be two phases for this project. The first phase is the "WE BEAT Group Wellness Education Program" and participants will be transitioned into the phase two HEART Club following phase one.

The trial will look at feasibility and acceptability of the program. Additional hypothesis include home whether exercise interventions can:

* be delivered without any associated serious cardiac events;
* will result in a decreased proportion of patients who are categorized as frail when compared to the cohort's pre-test baseline.
* will result in increased measured peak oxygen consumption when compared with their pre-intervention baseline.
* will result in increased step counts measured monthly from baseline to end of intervention
* will improve self-reported quality of life from baseline to post-intervention.
* will result in increased patient reported activity level from baseline to post-intervention

ELIGIBILITY:
Inclusion Criteria:

* Males and females with Fontan physiology who are 13 to <19 years of age at enrollment
* Own a mobile device capable of installing the University of Michigan Patient Portal application
* Fluent in English
* Participant consent or parental/guardian consent and participant assent

Exclusion Criteria:

* Height < 130 centimeters
* Current intravenous inotropic drugs
* Severe ventricular dysfunction assessed qualitatively by clinical echocardiography within six months prior to enrollment.
* Severe valvar regurgitation, ventricular outflow obstruction, or aortic arch obstruction assessed by clinical echocardiography within six months prior to enrollment.
* History of arrhythmia with exercise (excluding isolated supraventricular or ventricular ectopy without symptoms).
* Inability to complete exercise testing at baseline screening.
* Noncardiac medical, developmental, and/or social disorder that would prevent successful completion of planned study testing or would invalidate its results.
* Suicidality or homicidality in the past 6 months.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in the Connor-Davidson Resilience Scale 10 | baseline, 6 weeks
  This is a 10 item self-report rating scale 0 (not true at all) to 4 (true nearly all the time). The overall score range from 0 (no resilience) to 40 (high Resilience).
Change in the Lurz-Wilde pediatric frailty score | baseline (prior to home exercise start), after exercise program (6 months)
  The Lurz-Wilde Frailty score is the sum of points scored across 5 domains of physical and mental functioning (weakness, slowness, shrinkage, exhaustion, diminished physical activity). The maximum score is 10. If a patient accumulates > 5 points, they are considered frail. If a patient accumulates 4-5 points, they are considered pre-frail.

SECONDARY OUTCOMES:
Feasibility of the 2-phase intervention based on recruitment information - number of participants that are: approached, eligible, enrolled | up to approximately 18 months
Feasibility of the 2-phase intervention based on sociodemographic data including: self-reported race, ethnicity, household income, and education level of primary caregiver | up to approximately 18 months
Feasibility of the home exercise intervention program based on the number of adverse events (AEs) Categorized by relatedness to the intervention | 6 months
  * Not related: Accidents and injuries not related to exercise prescription, illnesses not attributed to cardiovascular status, Cardiac events that are not temporally related to prescribed exercise sessions
  * Possibly: Musculoskeletal complaints consistent with overuse or repetitive stress injury with a mechanism that is not consistent with the prescribed of exercise, Cardiac events/symptoms that occur between 90 to180 minutes after exercise
  * Probably: Musculoskeletal complaints consistent with overuse or repetitive stress injury that are consistent with the prescribed mechanism of exercise, Cardiac events/symptoms that occur between 15 minutes to 90 minutes after prescribed exercise
  * Definitely: Accidents or injuries that occur during prescribed exercise, Cardiac events/symptoms that occur during or up to 15 minutes after prescribed exercise
Change in the Patient Reported Outcome Measures Information System (PROMIS) pediatric physical activity -short form 4a | baseline (prior to home exercise start), after exercise program (6 months)
  This is a 4-item questionnaire that asks participants about their level of physical activity in the past 7 days. Items are scored on a 5-point scale. Scores range from 4 to 20 with 4 indicating low physical activity and 20 indicating high physical activity (better outcome).
Change in the Patient-Reported Outcomes Measurement Information System Pediatric Profile-25 2.0 (PROMIS-25) | baseline (prior to home exercise start), after exercise program (6 months)
  PROMIS-25 measures quality of life (i.e., depression, anxiety, and pain interference). The 25 items are on a 1-5 scale and are scored using the Health Measures Scoring Service with higher scores indicating a lower quality of life.
Seven day running average step counts | baseline (week 1 of exercise program), last week of exercise program (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hansen, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No